CLINICAL TRIAL: NCT00006942
Title: A Phase II Trial of Bryostatin in Combination With Cisplatin in Patients With Recurrent or Persistent Epithelial Ovarian Cancer
Brief Title: Bryostatin 1 and Cisplatin in Treating Patients With Advanced Recurrent or Residual Ovarian Epithelial, Fallopian Tube, or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02831; NCI-2012-02831 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PHII-21 (Other: City of Hope); T99-0039 (Other: CTEP); N01CM17101 (NIH)
Record Dates: First submitted 2000-12-06; First posted 2003-01-27 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2013-08

CONDITIONS: Fallopian Tube Cancer; Primary Peritoneal Cavity Cancer; Recurrent Ovarian Epithelial Cancer; Stage III Ovarian Epithelial Cancer; Stage IV Ovarian Epithelial Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Carcinoma, Ovarian Epithelial | interventions — bryostatin 1; Bryostatins; Cisplatin

ARMS (1):
- Treatment (bryostatin 1, cisplatin) (Experimental): Patients receive bryostatin 1 IV continuously over 72 hours immediately followed by cisplatin IV over 1 hour. Treatment continues every 3 weeks for a minimum of 2 courses in the absence of disease progression.
  Interventions: Drug: bryostatin 1; Drug: cisplatin; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: bryostatin 1 — Given IV
  Other Names: B705008K112; BRYO; Bryostatin
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase II trial to study the effectiveness of combining bryostatin 1 and cisplatin in treating patients who have advanced recurrent or residual ovarian epithelial, fallopian tube, or primary peritoneal cancer. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the overall response rate and the complete response rate of patients with platinum-refractory ovarian cancer who are treated with infusional Bryostatin-1 given in combination with intravenous cisplatin.

II. To estimate the duration of response in these patients. III. To obtain tissue in order to evaluate the molecular determinants of apoptosis including: p53 status, WAF1/CIP1 gene expression prior to and directly after chemotherapy, bcl-2 gene expression in vivo, bcl-2/bax ratio, p21, and the extent of apoptosis determined by the TdT assay; and the molecular determinants of DNA damage and repair including: expression levels of ERCC1.

OUTLINE: This is a multicenter study.

Patients receive bryostatin 1 IV continuously over 72 hours immediately followed by cisplatin IV over 1 hour. Treatment continues every 3 weeks for a minimum of 2 courses in the absence of disease progression.

Patients are followed for survival.

PROJECTED ACCRUAL: A total of 18-32 patients will be accrued for this study within 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Advanced recurrent or residual ovarian, fallopian tube, or papillary primary peritoneal cancer which has been histologically confirmed
* Eligible patients include patients with measurable disease who have progressed while on chemotherapeutic treatment, patients with biopsy-proven persistent, clinically-measurable disease with best response as stable at the completion of planned first-line therapy, patients with persistent or recurrent disease with rising CA-125 to levels at least twice normal; the CA-125 increase must be documented by two independent measurements; no patient may have received more than two prior regimens of chemotherapy including first-line treatment
* Patients must have a Karnofsky performance status of greater than or equal to 50% and an estimated survival of at least three months
* Measured or calculated clearance >= 60 ml/min
* AGC >= 1800/mm^3
* Plts >= 100,000/mm^3
* Bilirubin =< 1.5 mg/dl
* SGOT less than 2 x upper limit of normal
* Previous radiotherapy or chemotherapy must have been completed at least three weeks before treatment under this protocol
* Patients must have the ability to give voluntary informed consent and to comply with the treatment and required tests
* Because Bryostatin is of unknown teratogenic potential, women of childbearing potential must have a negative pregnancy test and must take adequate precautions to prevent pregnancy during treatment
* Patients with any non-malignant intercurrent illness (e.g. cardiovascular, pulmonary, or central nervous system disease) which is either poorly controlled with currently available treatment, or is of such severity that the investigators deem it unwise to enter the patient on protocol shall be ineligible
* Patients currently being treated for severe infection or who are recovering from major surgery are ineligible until recovery is deemed complete by the investigator
* The extent of all evaluable and nonevaluable disease must be documented; pretreatment radiographic examinations should be done no earlier than 4 weeks (28 days) prior to the first course of chemotherapy; pre-treatment chemistries and CA-125 levels should be done no earlier than two weeks (14 days) prior to initiation of chemotherapy; (in calculating days of tests and measurements, the day a test or measurement is done is considered day 0; therefore, if a test is done on Monday, the Monday four weeks later would be considered day 28; this allows for efficient patient scheduling without exceeding the guidelines)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2000-10; Primary Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Overall survival | Time from first day of treatment to time of death due to any cause, assessed up to 9 years
Progression-free survival | Time from first day of treatment to the first observation of disease progression or death due to any cause, assessed up to 9 years
Time to progression | Time from first day of treatment to the first observation of disease progression or death due to disease, assessed up to 9 years

SECONDARY OUTCOMES:
Response rate (CR or PR) | Up to 9 years
  Exact 95% confidence intervals will be calculated.
Time to treatment failure | Up to 9 years
  Estimated using the product-limit method of Kaplan and Meier.
Duration of response | Up to 9 years
  Estimated using the product-limit method of Kaplan and Meier.
Incidence by severity and type of toxicity based on the National Cancer Institute (NCI) Common Toxicity Criteria v2.0 and NCI Myalgia Toxicity Grading Scale | Up to 9 years
Association between p53, p21, bcl-2, bax, bcl-2/bax, ERCC-1, and Tdt and tumor response to chemotherapy (CR/PR vs not) | Prior to initiation of chemotherapy
  Proportions and Fisher's exact test will be used. Medians, ranges, quartiles and the Wilcoxon two-sample test will be used.
Association between p53, p21, bcl-2, bax, bcl-2/bax, ERCC-1, and Tdt and tumor response to chemotherapy (CR/PR vs not) | Day 5 of course 2
  Proportions and Fisher's exact test will be used. Medians, ranges, quartiles and the Wilcoxon two-sample test will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Morgan, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope, Duarte, California, United States